CLINICAL TRIAL: NCT01319331
Title: The Effects of Open Label Alpha-1 Antitrypsin on the Progression of Type 1 Diabetes in Subjects With Detectable C-peptide
Brief Title: The Effects of Alpha-1 Antitrypsin (AAT) on the Progression of Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Omni Bio Pharmaceutical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0667
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Type 1 Diabetes
Keywords: diabetes; type 1 diabetes; AAT; Alpha-1 Antitrypsin
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alpha-1 Antitrypsin (AAT, Aralast NP) (Experimental): Alpha-1 Antitrypsin (AAT, Aralast NP) as prescribed for study duration
  Interventions: Drug: Alpha 1-Antitrypsin (AAT, Aralast NP)

INTERVENTIONS:
Drug: Alpha 1-Antitrypsin (AAT, Aralast NP) — Eligible subjects will be treated once a week for 8 weeks (8 total treatments).
  Other Names: Alpha-1 Antitrypsin; AAT; Aralast NP

SUMMARY:
The purpose of this study is to determine if the drug Alpha-1 Antitrypsin (AAT, Aralast NP) will preserve beta-cell function and help slow the progression of type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes Mellitus based on ADA Criteria for fewer than 5 years but more than 100 days
* 6-45 years of age, inclusive. To assess safety, we will initially enroll 8 patients over the age of 16. Following the last infusion of the 8th patient, we will assess adverse events. As long as there are no stopping criteria met for these 8 patients we will decrease the age criteria down to 6 years old.
* C-peptide increase during screening mixed meal tolerance test with a minimal stimulated value of ≥ 0.2 pmol/mL.
* Positive for antibodies to insulin (if insulin autoantibody positive only, determination must be within two weeks of insulin initiation), GAD-65, IA-2 or ZnT8
* Agree to intensive management of diabetes with an HgbA1c goal of < 7.0%
* If female, (a) surgically sterile or (b) postmenopausal or (c) if of reproductive potential, willing to use medically acceptable birth control (e.g. female hormonal contraception, barrier methods or sterilization. ) until 3 months after completion of any treatment period
* If male and of reproductive potential, willing to use medically acceptable birth control until 3 months after completion of any treatment period, unless the female partner is postmenopausal or surgically sterile
* Serum creatinine ≤ 1.5 x upper limit of normal
* AST < 2 times the upper limit of normal
* Hematology:WBC > 3000 x 109/L; platelets > 100 x 109/L; hemoglobin > 10.0 g/dL.

Exclusion Criteria:

* Unable or unwilling to comply with the requirements of the study protocol
* Body Mass Index (BMI) > 30 kg/m2
* Unstable blood sugar control defined as one or more episodes of severe hypoglycemia (defined as hypoglycemia that required the assistance of another person) within the last 30 days
* Previous immunotherapy for T1D
* Administration of an experimental agent for T1D at any time or use of an experimental device for T1D within 30 days of screening, unless approved by the study PI
* History of any organ transplant, including islet cell transplant
* Active autoimmune or immune deficiency disorder (e.g. sarcoidosis, rheumatoid arthritis)
* Serum bilirubin > ULN, except those subjects whose abnormal values were attributed to any stable, benign condition (such as Gilbert's Syndrome) may be included
* TSH outside the normal range at screening, except those subjects on stable doses of thyroid hormone replacement therapy may be included
* Known HIV positivity, active hepatitis B or active hepatitis C infection
* Anticipated pregnancy during active dosing or within 3 months after completion of active dosing phase
* History of a malignant neoplasm within the previous 5 years (except in situ cervical cancer and curable non-melanoma skin malignancy)
* Any social condition or medical condition that would, in the opinion of the investigator, prevent complete participation in the study or that would pose a significant hazard to the subjects' participation
* History of active substance abuse within 12 months of screening
* A psychiatric or medical disorder that would prevent giving informed consent
* Individuals with a history of IgA deficiency
* Individuals with a history of hypersensitivity to AAT

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2015-10 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To assess participant safety & feasibility of study drug administration | Study duration is 2 years

SECONDARY OUTCOMES:
To assess AAT treatment on the maintenance of c-peptide production | Stimulated c-peptide at year one and two.
Assess the effects of AAT on glycemic variability and A1c. | Continuous Glucose Monitoring at one and two years.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Gottlieb, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center for Childhood Diabetes, Aurora, Colorado, United States

REFERENCES:
- [Derived] Ozeri E, Mizrahi M, Shahaf G, Lewis EC. alpha-1 antitrypsin promotes semimature, IL-10-producing and readily migrating tolerogenic dendritic cells. J Immunol. 2012 Jul 1;189(1):146-53. doi: 10.4049/jimmunol.1101340. Epub 2012 May 25. PMID 22634621
- See also: Related Info — http://www.barbaradaviscenter.org/